CLINICAL TRIAL: NCT05797792
Title: CHemical OptImization of Cerebral Embolectomy in Patients With Acute Stroke Treated With Mechanical Thrombectomy 2 (CHOICE 2 TRIAL)
Brief Title: CHemical OptImization of Cerebral Embolectomy 2 (CHOICE 2).
Acronym: CHOICE2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Angel Chamorro, M.D., Ph.D., Director, Comprehensive Stroke Center, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHOICE 2; 2023-504262-32 (EudraCT Number)
Record Dates: First submitted 2023-03-09; First posted 2023-04-04 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Stroke, Acute Ischemic; Stroke, Acute
Keywords: Mechanical Thrombectomy; Recanalization; Reperfusion; Alteplase
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, randomized, open, blinded end-point assessment phase III trial
Who Masked: Outcomes Assessor
Masking Description: The evaluation of the primary outcome measure (modified Rankin Scale Score 0-1 at day 90) will be conducted by central blinded evaluators following a structured questionnaire. The evaluation of imaging outcome measures will be conducted at the Imaging Central Core Laboratory by blinded evaluators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraarterial alteplase (Experimental): All the patients will be given a 15 minutes IA infusion of alteplase (Actylise®) at a drug concentration of 1.0 mg/ml. At 15 minutes of IA treatment onset, the infusion will be stopped and the angiographic score assessed. Study drug will be prepared according to the following steps: 1/ Dilute 2 vials of 10 mgs (rt-PA) in 20 cc of sterile water for injection (SWI), to attain a 20 ml solution at a concentration of 1mg/ml; 2. Calculate the volume of cc of infusion and therefore the total dose as per the formula: (Patient's weight in Kgs multiplied by 0.225). A patient of 89 Kgs or more will receive 20.0 cc of infusion for 15 min, totaling a dose of 20.0 mg of rt-PA.
  Interventions: Drug: Intraarterial alteplase
- No intervention (No Intervention): Patients allocated to this arm will receive a similar care to patients allocated to IA alteplase except the thrombolytic

INTERVENTIONS:
Drug: Intraarterial alteplase — See arm/group descriptions.
  Other Names: Intraarterial recombinant tissue plasminogen activator (rt-PA)
  Arms: Intraarterial alteplase

SUMMARY:
Multi-center, randomized, parallel-group, superiority study to compare the efficacy of adjunct intra-arterial rt-PA versus not adjunct intra-arterial rt-PA in the improvement of the efficacy of mechanical thrombectomy in patients with large vessel occlusion acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic large vessel occlusion (LVO) in the anterior circulation (ICA, ACA or MCA) treated with MT resulting in a mTICI score 2b/3 at end of the procedure. Patients with a mTICI score 2b/3 on the diagnostic cerebral angiography before the onset of MT are also eligible for the study.
* Estimated delay to onset of rescue intraarterial rt-PA administration <24 hours from symptom onset, defined as the point in time the patient was last seen well.
* No significant pre-stroke functional disability (modified Rankin scale 0-1), or mRS >1 that according to the investigator is not related to neurological disease (i.e., amputation, blindness)
* Age ≥18
* ASPECTS >6 on non-contrast CT (NCCT) scan if symptoms lasting <4.5 hours of last seen well. In patients with >4.5h of last seen well, a CT-perfusion (Flow maps) or MRI-perfusion should be considered instead of NCCT, especially if >9h have elapsed, or in seriously ill patients (i.e., NIHSS>17). Nonetheless, if a perfusion study is not available, NCCT can still be used as long as it is confirmed without a doubt that the ASPECTS is > 6.
* Informed consent, obtained from patient or acceptable patient surrogate, or Differed Informed Consent (DIC) to avoid any delay in the initiation of the mechanical thrombectomy and the i.a thrombolysis. The DIC will be signed by the patient or acceptable patient surrogate at any time after the tPA treatment is started.

Exclusion Criteria:

* NIHSS score on admission >25
* Contraindication to IV t-PA as per local national guidelines (except time to therapy)
* Use of carotid artery stents during the endovascular procedure requiring dual antiplatelet therapy during the first 24h
* Need of more than 3 passes (per vessel) or more than a total of 5 passes (in more than one vessel) to complete the endovascular procedure
* Female who is pregnant or lactating or has a positive pregnancy test at time of admission
* Current participation in another investigation drug or device treatment study
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
* Known coagulopathy, INR > 1.7
* Platelets < 50,000
* Renal Failure as defined by a serum creatinine > 3.0 mg/dl (or 265.2 μmol/l) or glomerular Filtration Rate [GFR] < 30
* Subject who requires hemodialysis or peritoneal dialysis, or who have a contraindication to an angiogram for whatever reason
* Any hemorrhage on CT/MRI
* Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT or MRI scan is normal
* Suspicion of aortic dissection
* Subject currently uses or has a recent history of illicit drug(s) or abuses alcohol
* History of life-threatening allergy (more than rash) to contrast medium
* SBP >185 mmHg or DBP >110 mmHg refractory to treatment
* Serious, advanced, terminal illness with anticipated life expectancy < 6 months
* Pre-existing neurological or psychiatric disease that would confound evaluation
* Presumed vasculitis or septic embolization
* Unlikely to be available for 90-day follow-up (i.e., no fixed home address, visitor from overseas)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-11-18 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale at day 90 | 90 days post treatment
  Proportion of patients with Modified Rankin Scale 0 or 1 at day 90 +/- 15d

SECONDARY OUTCOMES:
Microvascular hypoperfusion on follow-up brain CTP | 36±24hours post treatment
  Proportion of patients with abnormal microvascular hypoperfusion on CT Perfusion
Volume of hypoperfusion on brain CTP | at 36h±24h post treatment
  Volume of hypoperfusion on brain CTP
Infarct Expansion Ratio (IER): Final infarct to initial ischemic tissue volumes on brain CTP | 36±24hours post treatment
  Infarct Expansion Ratio (IER): Final infarct to initial ischemic tissue volumes on brain CTP at 36±24hours post MT.
Barthel Scale score | day 90 post treatment
  Barthel Scale score of 95 to 100, (min value 0, max value 100, higher score better outcome)
EuroQol Group 5-Dimension Self-Report Questionnaire (EQ-5D-3L) | day 90 post treatment
  Quality of life measured with the EuroQol Group 5-Dimension Self-Report Questionnaire (EQ-5D-3L) The score has five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Shift analysis of the modified Rankin Scale (mRS) | day 90 post treatment
  Shift analysis of the modified Rankin Scale (mRS), at day 90 (min value 0, max value 6, higher score worse outcome)

OTHER OUTCOMES:
SAFETY OUTCOME: Mortality at 90 days | Day 90
  Mortality at 90 days
SAFETY OUTCOME: symptomatic intracerebral hemorrahge (sICH ) rate at 24 hours. | 24hours post MT
  Symptomatic ICH will be classified as per the European Cooperative Acute Stroke Study (ECASS) 3 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Angel Chamorro, MD, PhD, Study Chair — Comprehensive Stroke Center, Hospital Clinic Barcelona; Arturo Renú, MD, PhD, Principal Investigator — Comprehensive Stroke Center, Hospital Clinic Barcelona; Juan F Arenillas, MD, Principal Investigator — Hospital Universitario de Valladolid; María del Mar Freijo, MD, Principal Investigator — Hospital Universitario de Cruces; Patricia de la Riva, MD, Principal Investigator — Hospital Donostia; M Dolores Fernándes, MD, Principal Investigator — Hospital Universitario de A Coruña; Pedro Vega, MD, Principal Investigator — Hospital Universitario Central de Asturias; Lluis Morales, MD, Principal Investigator — Hospital Universitario La Fe de Valencia; Laura Dorado, MD, Principal Investigator — Hospital Germans Trias i Pujol de Badalona; Mikel Terceño, MD, Principal Investigator — Hospital Universitario Dr. Josep Trueta de Girona; Ana Morales, MD, Principal Investigator — Hospital Universitario Virgen de Arrixaca Murcia; Maria Herrera, MD, Principal Investigator — Hospital of Navarra; Raquel Delgado, MD, Principal Investigator — Hospital Universitario Son Espases Mallorca; Nicolás López, MD, Principal Investigator — Hospital Universitario Dr. Balmis Alicante; Pol Camps, MD, Principal Investigator — Hospital Universitario de la Santa Creu i Sant Pau Barcelona
Locations (14):
- Spain (14):
  - Hospital Universitario de A Coruña, A Coruña, Spain
  - Hospital Universitario Dr. Balmis, Alicante, Spain
  - Hospital Germans Trías i Pujol, Badalona, Spain
  - Hospital Clinic Barcelona, Barcelona, Spain
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Spain
  - Hospital Universitario de Cruces, Bilbao, Spain
  - Hospital Josep Trueta, Girona, Spain
  - Hospital Universitario Virgen de la Arrixaca, Murcia, Spain
  - Hospital Universitario Central de Asturias, Oviedo, Spain
  - Hospital Universitario Son Espases, Palma de Mallorca, Spain
  - Hospital Universitario de Navarra, Pamplona, Spain
  - Hospital Universitario de Donostia, San Sebastián, Spain
  - Hospital Univesitario y Politénico La Fe, Valencia, Spain
  - Hospital Universitario de Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data on outcome measures will be published along with the main results of the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available after publication of main study results.
Access Criteria: The IPD will be available from the Sponsor of the trial on reasonable request.

REFERENCES:
- [Background] Chamorro A, Blasco J, Lopez A, Amaro S, Roman LS, Llull L, Renu A, Rudilosso S, Laredo C, Obach V, Urra X, Planas AM, Leira EC, Macho J. Complete reperfusion is required for maximal benefits of mechanical thrombectomy in stroke patients. Sci Rep. 2017 Sep 14;7(1):11636. doi: 10.1038/s41598-017-11946-y. PMID 28912596
- [Background] Davalos A, Cobo E, Molina CA, Chamorro A, de Miquel MA, Roman LS, Serena J, Lopez-Cancio E, Ribo M, Millan M, Urra X, Cardona P, Tomasello A, Castano C, Blasco J, Aja L, Rubiera M, Gomis M, Renu A, Lara B, Marti-Fabregas J, Jankowitz B, Cerda N, Jovin TG; REVASCAT Trial Investigators. Safety and efficacy of thrombectomy in acute ischaemic stroke (REVASCAT): 1-year follow-up of a randomised open-label trial. Lancet Neurol. 2017 May;16(5):369-376. doi: 10.1016/S1474-4422(17)30047-9. Epub 2017 Mar 16. PMID 28318984
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Background] Renu A, Blasco J, Millan M, Marti-Fabregas J, Cardona P, Oleaga L, Macho J, Molina C, Roquer J, Amaro S, Davalos A, Zarco F, Laredo C, Tomasello A, Guimaraens L, Barranco R, Castano C, Vivas E, Ramos A, Lopez-Rueda A, Urra X, Muchada M, Cuadrado-Godia E, Camps-Renom P, Roman LS, Rios J, Leira EC, Jovin T, Torres F, Chamorro A; CHOICE Investigators. The Chemical Optimization of Cerebral Embolectomy trial: Study protocol. Int J Stroke. 2021 Jan;16(1):110-116. doi: 10.1177/1747493019895656. Epub 2019 Dec 18. PMID 31852410
- [Background] Renu A, Millan M, San Roman L, Blasco J, Marti-Fabregas J, Terceno M, Amaro S, Serena J, Urra X, Laredo C, Barranco R, Camps-Renom P, Zarco F, Oleaga L, Cardona P, Castano C, Macho J, Cuadrado-Godia E, Vivas E, Lopez-Rueda A, Guimaraens L, Ramos-Pachon A, Roquer J, Muchada M, Tomasello A, Davalos A, Torres F, Chamorro A; CHOICE Investigators. Effect of Intra-arterial Alteplase vs Placebo Following Successful Thrombectomy on Functional Outcomes in Patients With Large Vessel Occlusion Acute Ischemic Stroke: The CHOICE Randomized Clinical Trial. JAMA. 2022 Mar 1;327(9):826-835. doi: 10.1001/jama.2022.1645. PMID 35143603
- [Background] Laredo C, Rodriguez A, Oleaga L, Hernandez-Perez M, Renu A, Puig J, Roman LS, Planas AM, Urra X, Chamorro A. Adjunct Thrombolysis Enhances Brain Reperfusion following Successful Thrombectomy. Ann Neurol. 2022 Nov;92(5):860-870. doi: 10.1002/ana.26474. Epub 2022 Aug 23. PMID 36054449
- [Background] Chamorro A, Torres F. Intra-arterial Alteplase vs Placebo After Successful Thrombectomy and Functional Outcomes in Patients With Large Vessel Occlusion Acute Ischemic Stroke-Reply. JAMA. 2022 Jun 28;327(24):2456. doi: 10.1001/jama.2022.7430. No abstract available. PMID 35763000